CLINICAL TRIAL: NCT01279720
Title: Phase I Gene Therapy Protocol for Adenosine Deaminase Deficiency
Brief Title: Gene Therapy ADA Deficiency
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03MI14
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2015-09-14 (Estimated); Status verified 2015-09

CONDITIONS: Adenosine Deaminase Deficiency
Keywords: Adenosine deaminase deficiency; Gene therapy
MeSH Terms: conditions — Severe combined immunodeficiency due to adenosine deaminase deficiency

ARMS (1):
- Intravenous infusion of transduced cells (Experimental): Intravenous infusion of transduced cells
  Interventions: Biological: Intravenous infusion of transduced cells

INTERVENTIONS:
Biological: Intravenous infusion of transduced cells — Intravenous infusion of transduced cells

SUMMARY:
Adenosine deaminase deficiency is an inherited disorder that results in severe abnormalities of the immune system and leaves children unable to fight infection. This trial aims to treat adenosine deaminase deficiency patients using gene therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who lack a human leukocyte antigen (HLA)-genotypically identical bone marrow donor OR phenotypically matched family or unrelated donor AND who show incomplete immune reconstitution on Polyethylene glycol-modified adenosine deaminase (PEG-ADA) enzyme replacement therapy (defined by absolute CD4+ count <300 cell/mm3 and who remain on immunoglobulin replacement therapy)
2. Diagnosis of ADA-SCID (Severe combined immunodeficiency (SCID) due to adenosine deaminase (ADA)confirmed by DNA sequencing OR by confirmed absence of <3% of ADA enzymatic activity in peripheral blood or (for neonates) in umbilical cord blood erythrocytes and/or leukocytes or in cultured fetal cells derived from either chorionic villus biopsy or amniocentesis, prior to institution of PEG-ADA replacement therapy
3. Parental/guardian/patient signed informed consent

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2003-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Immunological reconstitution | 5 years
  Measurement of Immunological reconstitution and Metabolic Correction. 5 year follow up of the last patient enrolled into study

SECONDARY OUTCOMES:
Incidence of adverse reactions | 5 years
  Incidence of adverse reactions. 5 year follow up of the last patient enrolled into study
Molecular characterisation of gene transfer | 5 years
  Molecular characterisation of gene transfer. 5 year follow up of the last patient enrolled into study
Normalisation of nutritional status, growth, and development | 5 years
  Normalisation of nutritional status, growth, and development. 5 year follow up of the last patient enrolled into study

CONTACTS AND LOCATIONS:
Locations (1):
- Great Ormond Street Hospital for Children NHS Trust, London, United Kingdom

REFERENCES:
- [Background] Aiuti A, Slavin S, Aker M, Ficara F, Deola S, Mortellaro A, Morecki S, Andolfi G, Tabucchi A, Carlucci F, Marinello E, Cattaneo F, Vai S, Servida P, Miniero R, Roncarolo MG, Bordignon C. Correction of ADA-SCID by stem cell gene therapy combined with nonmyeloablative conditioning. Science. 2002 Jun 28;296(5577):2410-3. doi: 10.1126/science.1070104. PMID 12089448
- [Background] Hoogerbrugge PM, van Beusechem VW, Fischer A, Debree M, le Deist F, Perignon JL, Morgan G, Gaspar B, Fairbanks LD, Skeoch CH, Moseley A, Harvey M, Levinsky RJ, Valerio D. Bone marrow gene transfer in three patients with adenosine deaminase deficiency. Gene Ther. 1996 Feb;3(2):179-83. PMID 8867866
- [Background] Hershfield MS. PEG-ADA: an alternative to haploidentical bone marrow transplantation and an adjunct to gene therapy for adenosine deaminase deficiency. Hum Mutat. 1995;5(2):107-12. doi: 10.1002/humu.1380050202. PMID 7749407